CLINICAL TRIAL: NCT03669640
Title: Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Effects of RO6889450 (Ralmitaront) in Patients With Schizophrenia or Schizoaffective Disorder and Negative Symptoms
Brief Title: A Study to Assess the Effects of RO6889450 (Ralmitaront) in Participants With Schizophrenia or Schizoaffective Disorder and Negative Symptoms
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was discontinued due to an interim analysis which indicated that ralmitaront was unlikely to meet its primary endpoint.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP40283
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia, Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Monotherapy (Experimental): Participants will receive RO6889450 or a dose-matched placebo. NOTE: Part A has completed enrollment.
  Interventions: Drug: RO6889450; Drug: Placebo
- Part B: Add-On Therapy (Experimental): Participants will receive a low or high dose of RO6889450 or a dose-matched placebo in addition to their usual anti-psychotic treatment(s).
  Interventions: Drug: RO6889450; Drug: Placebo

INTERVENTIONS:
Drug: RO6889450 — Participants will receive a once-daily, oral dose of RO6889450 for 12 weeks.
Drug: Placebo — Participants will receive a once-daily, oral dose of placebo matched to RO6889450 for 12 weeks.

SUMMARY:
This study investigates the effects of RO6889450 on the negative symptoms associated with schizophrenia and schizoaffective disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnosis of schizophrenia or schizoaffective disorder as confirmed by the Mini International Neuropsychiatric Interview (MINI)
* Part B only: Stable treatment with a dopamine/serotonin (D2/5HT2A) antagonist or pure D2 antagonist(s), or a D2 partial agonist for a minimum of 6 months and receiving no more than two antipsychotics
* Medically stable during the 3 months prior to study entry
* Participant is an outpatient with no psychiatric hospitalizations within the prior 6 months
* PANSS negative symptom factor score of 18 or higher
* The following rating on items of the PANSS: (a) less than 5 on G8 (uncooperativeness), P1 (delusions), P3 (hallucinations), P4 (excitement/hyperactivity), and P6 (suspiciousness/persecution); (b) less than 4 on P7 (hostility), and G14 (poor impulse control)
* Has an informant who is considered reliable by the Investigator
* Body mass index (BMI) between 18-40 kg/m2 inclusive
* Female participants are eligible to participate if not pregnant, not breastfeeding and agree to remain abstinent or use acceptable contraceptive methods during the treatment period and for at least 28 days after the last dose of study drug

Exclusion Criteria:

* Moderate to severe substance use disorder within six months of study entry (excluding nicotine or caffeine) as defined by DSM-5
* Extrapyramidal symptom rating scale (ESRS-A CGI) subscore greater than or equal to 3
* Other current DSM-5 diagnosis (e.g., bipolar disorder, major depressive disorder)
* PANSS item G6 (depression) greater than or equal to 5
* Significant risk of suicide or harming him- or herself or others according to the Investigator's judgment
* A prior or current general medical condition that might be impairing cognition or other psychiatric functioning
* Positive result at screening for hepatitis B surface antigen (HBsAg), hepatitis C (HCV), or HIV-1 and HIV-2. HCV antibody positive participants are eligible if HCV RNA is negative
* Tardive dyskinesia that is moderate to severe or requires treatment
* History of neuroleptic malignant syndrome
* Average triplicate Fridericia's Correction Formula (QTcF) interval greater than 450 milliseconds (msec) for males and 470 msec for females or other clinically significant abnormality on screening electrocardiogram (ECG) based on centralized reading
* Clinically significant abnormalities in laboratory safety test results
* Significant or unstable physical condition that in the investigator's judgment might require a change in medication or hospitalization during the course of the study
* On more than one antidepressant, or if on one antidepressant, a change in dose within 28 days prior to screening
* History of clozapine treatment
* History of treatment with electroconvulsive therapy (ECT)
* Concomitant use of prohibited medications
* Positive urine drug screen for amphetamines, methamphetamines, opiates, buprenomorphine, methadone, cannabinoids, cocaine, and barbiturates
* Receipt of an investigational drug within 28 days or five times the half-life of the investigational drug (whichever is longer) before the first study drug administration
* Donation of blood over 400 mL within 3 months prior to screening
* Diagnosis of COVID-19 infection (confirmed or presumptive) 4 weeks prior to screening or during screening. Participants can be re-screened after 4 weeks of full recovery in addition to Investigator and/or institutional approval to enroll

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 131 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (45):
- United States (28):
  - CITrials, Inc., Bellflower, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - California Clinical Trials, Glendale, California
  - Synergy San Diego, Lemon Grove, California
  - Catalina Research Institute LLC - MRA, Montclair, California
  - CITrials, Inc., Riverside, California
  - California Neuropsychopharmacology Clinical Research Institute, LLC, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - Collaborative Neuroscience Network Inc., Torrance, California
  - Yale School of Medicine - CT Mental Health Center (CMHC) - Schizophrenia Research Clinic, New Haven, Connecticut
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Lifestream Behavioral Center, Leesburg, Florida
  - Advanced Research Institute of Miami, Miami, Florida
  - Health Synergy Clinical Research, Okeechobee, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - CBH Health, Gaithersburg, Maryland
  - Precise Research Centers, Flowood, Mississippi
  - Psych Care Consultants Research, St Louis, Missouri
  - Millennium Psychiatric Associates, LLC, St Louis, Missouri
  - Manhattan Psychiatric Center; Psychopharmacology Research Unit, New York, New York
  - JPS Health Network, Fort Worth, Texas
  - Pillar Clinical Research LLC, Garland, Texas
  - Baylor College of Medicine, Houston, Texas
  - University Hills Clinical Research, Irving, Texas
  - The Solace Center, Missouri City, Texas
  - Psychiatry & Behavioral Center, Richmond, Texas
  - @ Health Texas, Richmond, Texas
- Japan (5):
  - Kohnodai Hp., National Center for Global Health and Medicine, Chiba
  - National Hospital Organization Ryukyu Hospital, Kunigami
  - National Center of Neurology and Psychiatry, Tokyo
  - Seishinkai Okehazama Hospital Fujita Kokoro Care Center, Toyoake
  - Hiyoshi Hospital, Yokohama
- Spain (5):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - Hosp Univ Fundacion Alcorcon, Madrid
  - Complejo Asistencial Universitario de Salamanca ? H. Clinico, Salamanca
- Ukraine (7):
  - CNCE Regional Clinical Psychiatric Hospital of Kirovohrad Regional Council, Nove, Katerynoslav Governorate
  - Communal Non-Commercial Enterprise of Kharkiv RC Regional clinical psychiatric hospital #3, Kharkiv, Kharkiv Governorate
  - Public NPE Kherson Regional Institution of Mental Care of Kherson RC, Kherson, Kherson Governorate
  - Municipal Non-Commercial Enterprise Odesa RMC for Mental Health of Odessa Regional Council, Odesa, Kherson Governorate
  - ME Dnipropetrovsk Regional Clinical Hospital n.a. I.I Mechnykov Dnipropetrovsk Regional Council, Dnipro, KIEV Governorate
  - Zakarpattia Regional Clinical Hospital n.a. Andrii Novak, Uzhhorod, KIEV Governorate
  - Communal NPE Vinnytsia Reg. Clin. Psychoneurolog. Hosp. n.a. O.I. Yushchenko of Vinnytsia RC, Vinnytsia, Podolia Governorate

REFERENCES:
- [Derived] Halff EF, Rutigliano G, Garcia-Hidalgo A, Howes OD. Trace amine-associated receptor 1 (TAAR1) agonism as a new treatment strategy for schizophrenia and related disorders. Trends Neurosci. 2023 Jan;46(1):60-74. doi: 10.1016/j.tins.2022.10.010. Epub 2022 Nov 8. PMID 36369028

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Monotherapy (Placebo): Participants received placebo each day (QD) for 12 weeks after a 1-week washout from their usual antipsychotic therapy.
- Part A: Monotherapy (150 mg): Participants received 150 mg of ralmitaront QD for 12 weeks after a 1-week washout from their usual antipsychotic therapy.
- Part B: Add-on Therapy (Placebo): Participants received placebo QD for 12 weeks in addition to their usual antipsychotic therapy.
- Part B: Add-on Therapy (45 mg): Participants received 45 mg of ralmitaront QD 12 weeks in addition to their usual antipsychotic therapy (prior to protocol v5; arm was removed thereafter).
- Part B: Add-on Therapy (150 mg): Participants received 150 mg of ralmitaront QD 12 weeks in addition to their usual antipsychotic therapy.
- Part B: Add-on Therapy (300 mg): Participants received 300 mg of ralmitaront QD 12 weeks in addition to their usual antipsychotic therapy (after protocol v5).
Period: Overall Study
Arm/Group | Part A: Monotherapy (Placebo) | Part A: Monotherapy (150 mg) | Part B: Add-on Therapy (Placebo) | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
Started | 15 | 12 | 37 | 5 | 30 | 32
Completed | 10 | 7 | 33 | 5 | 27 | 29
Not Completed | 5 | 5 | 4 | 0 | 3 | 3
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0 | 1 | 3
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Disease Relapse | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Monotherapy (Placebo) | Part A: Monotherapy (150 mg) | Part B: Add-on Therapy (Placebo) | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg) | Total
Number analyzed (Participants) | 15 | 12 | 37 | 5 | 30 | 32 | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (9.9) | 43.3 (6.6) | 41.3 (9.7) | 41.6 (11.3) | 40.0 (9.6) | 40.9 (9.2) | 41.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 10 | 0 | 11 | 12 | 39
  Male | 12 | 9 | 27 | 5 | 19 | 20 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 0 | 6 | 5 | 14
  Not Hispanic or Latino | 14 | 11 | 35 | 5 | 24 | 27 | 116
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 8 | 0 | 6 | 4 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 12 | 9 | 11 | 5 | 7 | 10 | 54
  White | 2 | 3 | 16 | 0 | 16 | 18 | 55
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Brief Negative Symptoms Scale (BNSS) Avolition/Apathy Subscore and Total Score at Baseline and Week 12
Description: The BNSS is a 13-item instrument designed for clinical trials that measures the severity of the negative symptoms of schizophrenia in five domains. There are 13 items organized into 6 subscales (anhedonia, distress, asociality, avolition, blunted affect, and alogia), each rated on a 7-point scale (0-6) where 0 = absent symptoms and 6 = severe symptoms. The total score is calculated by summing the individual items (13) of each subscale and has a range of 0-78. The avolition/apathy subscale contains 2 items with a total score range of 0-12.
Time Frame: Baseline to Week 12
Population: The modified intent-to-treat (mITT) population included all randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part A: Monotherapy (Placebo) | Part A: Monotherapy (150 mg) | Part B: Add-on Therapy (Placebo) | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
Number analyzed (Participants) | 15 | 12 | 37 | 5 | 30 | 32
Units on a scale
  Baseline Avolition/Apathy Subscore: number analyzed (Participants) | 14 | 12 | 36 | 5 | 29 | 32
  Baseline Avolition/Apathy Subscore | 5.71 (2.81) | 5.50 (2.71) | 6.0 (2.3) | 6.2 (1.3) | 5.8 (1.9) | 5.9 (2.4)
  Week 12 (Day 84) Avolition/Apathy Subscore: number analyzed (Participants) | 10 | 6 | 31 | 4 | 20 | 21
  Week 12 (Day 84) Avolition/Apathy Subscore | 5.50 (2.55) | 4.67 (3.27) | 5.0 (1.9) | 5.3 (1.0) | 4.1 (2.1) | 4.7 (2.1)

2. Secondary Outcome: Clinical Global Impression Severity (CGI-S) Overall Scores
Description: The CGI-S is an absolute measure assessing how mentally ill the participant is at the time of the assessment on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). On the scale, the value 0 corresponds to 'not assessed', which will be excluded from the analyses. The values 1 to 7 will be transformed into the 0 to 6 range prior to statistical analysis for the question on the measure ("Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?"), making the total score range 0-6.
Time Frame: Baseline to week 12
Population: The modified intent-to-treat (mITT) population included all randomized participants who received at least one dose of study drug. Data for this endpoint was not collected for Part B on Day 70.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part A: Monotherapy (Placebo) | Part A: Monotherapy (150 mg) | Part B: Add-on Therapy (Placebo) | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
Number analyzed (Participants) | 15 | 12 | 37 | 5 | 30 | 32
Units on a scale
  Baseline | 3.600 (0.507) | 3.667 (0.492) | 4.1 (0.7) | 3.8 (0.4) | 3.9 (0.7) | 4.0 (0.7)
  Day 14: number analyzed (Participants) | 15 | 10 | 35 | 4 | 27 | 31
  Day 14 | 3.467 (0.516) | 3.700 (0.483) | 4.0 (0.6) | 3.8 (0.5) | 3.8 (0.6) | 4.0 (0.8)
  Day 28: number analyzed (Participants) | 10 | 9 | 34 | 4 | 26 | 29
  Day 28 | 3.500 (0.527) | 3.333 (0.500) | 3.9 (0.8) | 3.8 (0.5) | 3.8 (0.6) | 3.7 (0.7)
  Day 42: number analyzed (Participants) | 11 | 8 | 32 | 4 | 24 | 26
  Day 42 | 3.636 (0.809) | 3.375 (0.744) | 3.8 (0.8) | 3.8 (0.5) | 3.6 (0.6) | 3.6 (0.7)
  Day 56: number analyzed (Participants) | 11 | 7 | 33 | 4 | 24 | 25
  Day 56 | 3.636 (0.505) | 3.143 (0.378) | 3.8 (0.8) | 3.8 (0.5) | 3.5 (0.7) | 3.5 (0.8)
  Day 70: number analyzed (Participants) | 10 | 7 | 0 | 0 | 0 | 0
  Day 70 | 3.500 (0.707) | 3.143 (0.690) |  |  |  |
  Day 84: number analyzed (Participants) | 10 | 6 | 31 | 4 | 20 | 22
  Day 84 | 3.700 (0.483) | 3.000 (0.632) | 3.7 (0.8) | 3.8 (0.5) | 3.4 (0.6) | 3.5 (0.7)

3. Secondary Outcome: CGI-S Negative Symptoms (NS) Scores
Description: The CGI-S-NS is similar to the CGI-S and is assessed on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). On the scale, the value 0 corresponds to 'not assessed', which will be excluded from the analyses. The values 1 to 7 will be transformed into the 0 to 6 range prior to statistical analysis for the question on the measure, making the total score range 0-6.
Time Frame: Baseline to week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part A: Monotherapy (Placebo) | Part A: Monotherapy (150 mg) | Part B: Add-on Therapy (Placebo) | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
Number analyzed (Participants) | 15 | 12 | 37 | 5 | 30 | 32
Units on a scale
  Baseline | 3.867 (0.743) | 3.917 (0.669) | 4.4 (0.6) | 4.2 (0.4) | 4.3 (0.7) | 4.3 (0.7)
  Day 14: number analyzed (Participants) | 15 | 10 | 35 | 4 | 27 | 31
  Day 14 | 3.600 (0.632) | 3.800 (0.632) | 4.3 (0.7) | 4.3 (0.5) | 3.9 (0.7) | 4.1 (0.7)
  Day 28: number analyzed (Participants) | 10 | 9 | 34 | 4 | 26 | 29
  Day 28 | 3.800 (0.632) | 3.778 (0.667) | 4.1 (0.8) | 4.3 (0.5) | 3.8 (0.7) | 3.9 (0.7)
  Day 42: number analyzed (Participants) | 11 | 8 | 32 | 4 | 24 | 26
  Day 42 | 3.727 (0.467) | 3.625 (0.518) | 3.9 (0.9) | 4.0 (0.0) | 3.8 (0.7) | 3.7 (0.7)
  Day 56: number analyzed (Participants) | 11 | 7 | 33 | 4 | 24 | 25
  Day 56 | 3.636 (0.674) | 3.714 (0.756) | 3.9 (0.8) | 4.0 (0.0) | 3.6 (0.7) | 3.5 (0.7)
  Day 70: number analyzed (Participants) | 10 | 7 | 0 | 0 | 0 | 0
  Day 70 | 3.500 (0.527) | 3.286 (0.756) |  |  |  |
  Day 84: number analyzed (Participants) | 10 | 6 | 31 | 4 | 20 | 22
  Day 84 | 3.400 (0.516) | 3.167 (0.753) | 3.9 (0.8) | 3.8 (0.5) | 3.4 (0.6) | 3.5 (0.9)

4. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Overall Scores
Description: The CGI-I assesses how much the participant's condition has changed at the time of the assessment in comparison to their condition at baseline. It uses a 7-point scale ranging from 1 (very much improved) to 7 (very much worse), where the value 0 corresponds to 'not assessed' and will be excluded from any analyses.
Time Frame: Up to Week 12 (Day 84)
Population: The modified intent-to-treat (mITT) population included all randomized participants who received at least one dose of study drug. Data for this endpoint was not collected for Part B Days 21, 35, and 70.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part A: Monotherapy (Placebo) | Part A: Monotherapy (150 mg) | Part B: Add-on Therapy (Placebo) | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
Number analyzed (Participants) | 15 | 12 | 37 | 5 | 30 | 32
Units on a scale
  Day 14: number analyzed (Participants) | 14 | 9 | 35 | 4 | 27 | 31
  Day 14 | 3.71 (0.91) | 3.56 (0.53) | 3.7 (0.4) | 4.0 (0.0) | 3.6 (0.5) | 3.6 (0.6)
  Day 21: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0
  Day 21 | 4.00 (NA) — SD cannot be calculated with a single value | 2.00 (NA) — SD cannot be calculated with a single value |  |  |  |
  Day 28: number analyzed (Participants) | 9 | 8 | 34 | 4 | 26 | 29
  Day 28 | 3.56 (0.73) | 3.50 (0.76) | 3.5 (0.7) | 4.0 (0.0) | 3.5 (0.8) | 3.4 (0.8)
  Day 35: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 0
  Day 35 | 3.50 (0.71) |  |  |  |  |
  Day 42: number analyzed (Participants) | 11 | 7 | 32 | 4 | 24 | 26
  Day 42 | 3.73 (0.65) | 3.29 (0.76) | 3.4 (0.7) | 3.8 (0.5) | 3.3 (0.8) | 3.3 (0.9)
  Day 56: number analyzed (Participants) | 10 | 7 | 33 | 4 | 24 | 25
  Day 56 | 3.70 (0.48) | 3.14 (0.69) | 3.4 (0.7) | 3.8 (0.5) | 3.4 (0.9) | 3.1 (1.0)
  Day 70: number analyzed (Participants) | 10 | 7 | 0 | 0 | 0 | 0
  Day 70 | 3.50 (0.71) | 2.86 (0.90) |  |  |  |
  Day 84: number analyzed (Participants) | 10 | 6 | 31 | 4 | 20 | 22
  Day 84 | 3.80 (0.42) | 3.00 (0.63) | 3.2 (0.7) | 3.8 (0.5) | 3.0 (0.9) | 3.0 (1.0)

5. Secondary Outcome: CGI-I Negative Symptoms Scores
Description: The CGI-I NS is similar to the CGI-I and assesses how much the participant's condition has changed at the time of the assessment in comparison to their condition at baseline. It uses a 7-point scale, where:
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse
Time Frame: Up to Week 12 (Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part A: Monotherapy (Placebo) | Part A: Monotherapy (150 mg) | Part B: Add-on Therapy (Placebo) | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
Number analyzed (Participants) | 15 | 12 | 37 | 5 | 30 | 32
Units on a scale
  Day 14: number analyzed (Participants) | 14 | 9 | 35 | 4 | 27 | 31
  Day 14 | 3.71 (0.61) | 3.44 (0.73) | 3.7 (0.5) | 4.0 (0.0) | 3.5 (0.6) | 3.5 (0.6)
  Day 21: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0
  Day 21 | 5.00 (NA) — SD cannot be calculated with a single value | 4.00 (NA) — SD cannot be calculated with a single value |  |  |  |
  Day 28: number analyzed (Participants) | 9 | 8 | 34 | 4 | 26 | 29
  Day 28 | 3.44 (0.73) | 3.38 (0.74) | 3.5 (0.7) | 4.0 (0.0) | 3.3 (0.7) | 3.2 (0.8)
  Day 35: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 0
  Day 35 | 4.50 (0.71) |  |  |  |  |
  Day 42: number analyzed (Participants) | 11 | 7 | 32 | 4 | 24 | 26
  Day 42 | 3.45 (0.69) | 3.43 (0.79) | 3.3 (0.6) | 3.5 (0.6) | 3.3 (0.8) | 3.2 (0.8)
  Day 56: number analyzed (Participants) | 10 | 7 | 33 | 4 | 24 | 25
  Day 56 | 3.50 (0.71) | 3.43 (0.53) | 3.2 (0.7) | 3.5 (0.6) | 3.2 (0.8) | 2.9 (0.8)
  Day 70: number analyzed (Participants) | 10 | 7 | 0 | 0 | 0 | 0
  Day 70 | 3.40 (0.70) | 3.00 (0.82) |  |  |  |
  Day 84: number analyzed (Participants) | 10 | 6 | 31 | 4 | 20 | 22
  Day 84 | 3.10 (0.74) | 2.83 (0.41) | 3.1 (0.7) | 3.0 (0.8) | 2.9 (0.9) | 2.8 (0.9)

6. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) Total Scores
Description: The PANSS Marder factors examine schizophrenia symptoms in five domains: positive symptoms, negative symptoms, disorganized thought, uncontrolled hostility/excitement, and depression/anxiety. The Marder factor positive symptom score (range = 8-56) measures responses to 8 items (P1,P3,P5,P6,N7,G1,G9,G12) while the negative symptom factor score (range = 7-49) consists of 7 items (N1,N2,N3,N4,N6,G7,G16). Each item is scored on a scale of 1-7, where 1 = an absence of symptoms and 7 = extreme symptoms. The positive and negative syndrome scale total score is the sum of the scores from each domain (range = 15-105); higher scores indicate greater severity of symptoms.
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part A: Monotherapy (Placebo) | Part A: Monotherapy (150 mg) | Part B: Add-on Therapy (Placebo) | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
Number analyzed (Participants) | 15 | 12 | 37 | 5 | 30 | 32
Units on a scale
  Baseline: number analyzed (Participants) | 14 | 12 | 37 | 5 | 30 | 32
  Baseline | 67.43 (9.35) | 67.92 (10.86) | 71.4 (10.3) | 62.8 (6.7) | 69.6 (11.1) | 67.8 (11.1)
  Day 14: number analyzed (Participants) | 13 | 10 | 36 | 4 | 26 | 30
  Day 14 | 68.38 (10.37) | 69.00 (11.40) | 67.3 (8.5) | 69.5 (13.5) | 67.4 (10.5) | 67.9 (13.6)
  Day 28: number analyzed (Participants) | 10 | 9 | 33 | 3 | 26 | 28
  Day 28 | 66.10 (10.38) | 65.44 (7.30) | 67.0 (10.9) | 81.3 (4.7) | 66.8 (11.4) | 66.5 (11.1)
  Day 42: number analyzed (Participants) | 11 | 8 | 32 | 4 | 24 | 24
  Day 42 | 70.09 (10.88) | 65.88 (12.01) | 68.3 (12.7) | 73.3 (9.8) | 61.8 (10.9) | 64.1 (12.5)
  Day 56: number analyzed (Participants) | 10 | 7 | 32 | 4 | 24 | 23
  Day 56 | 66.60 (8.13) | 61.14 (6.91) | 64.3 (11.7) | 70.0 (7.1) | 63.2 (14.4) | 61.4 (11.7)
  Day 70: number analyzed (Participants) | 10 | 7 | 0 | 0 | 0 | 0
  Day 70 | 68.50 (7.65) | 59.57 (7.14) |  |  |  |
  Day 84 (Week 12): number analyzed (Participants) | 10 | 6 | 31 | 4 | 20 | 21
  Day 84 (Week 12) | 64.70 (13.92) | 59.17 (6.27) | 64.4 (12.2) | 74.8 (7.2) | 59.0 (11.1) | 60.9 (11.3)

7. Secondary Outcome: PANSS Symptom Factor Scores
Description: The PANSS Marder factors examine schizophrenia symptoms in five domains: positive symptoms, negative symptoms, disorganized thought, uncontrolled hostility/excitement, and depression/anxiety. The Marder factor positive symptom score (range = 8-56) measures responses to 8 items (P1,P3,P5,P6,N7,G1,G9,G12) while the negative symptom factor score (range = 7-49) consists of 7 items (N1,N2,N3,N4,N6,G7,G16). Each item is scored on a scale of 1-7, where 1 = an absence of symptoms and 7 = extreme symptoms.
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part A: Monotherapy (Placebo) | Part A: Monotherapy (150 mg) | Part B: Add-on Therapy (Placebo) | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
Number analyzed (Participants) | 15 | 12 | 37 | 5 | 30 | 32
Units on a scale
  Baseline - Negative symptoms: number analyzed (Participants) | 14 | 12 | 37 | 5 | 30 | 32
  Baseline - Negative symptoms | 21.29 (4.45) | 21.00 (5.20) | 23.0 (4.7) | 20.6 (3.3) | 23.3 (4.7) | 23.5 (4.1)
  Day 14 - Negative symptoms: number analyzed (Participants) | 13 | 10 | 36 | 4 | 26 | 30
  Day 14 - Negative symptoms | 22.46 (5.13) | 20.40 (3.95) | 22.9 (3.4) | 20.8 (2.9) | 21.8 (4.5) | 22.2 (5.3)
  Day 28 - Negative symptoms: number analyzed (Participants) | 10 | 9 | 33 | 3 | 26 | 28
  Day 28 - Negative symptoms | 18.40 (6.67) | 20.44 (3.68) | 20.9 (4.8) | 20.3 (3.1) | 21.5 (4.0) | 22.1 (4.9)
  Day 42 - Negative symptoms: number analyzed (Participants) | 11 | 8 | 32 | 4 | 24 | 24
  Day 42 - Negative symptoms | 21.09 (5.45) | 19.00 (5.50) | 21.3 (4.5) | 22.3 (3.2) | 21.5 (5.1) | 20.7 (5.1)
  Day 56 - Negative symptoms: number analyzed (Participants) | 10 | 7 | 32 | 4 | 24 | 23
  Day 56 - Negative symptoms | 21.10 (5.93) | 18.71 (4.72) | 20.4 (4.7) | 21.8 (4.2) | 19.8 (4.9) | 20.3 (5.7)
  Day 70 - Negative symptoms: number analyzed (Participants) | 10 | 7 | 0 | 0 | 0 | 0
  Day 70 - Negative symptoms | 21.20 (5.07) | 17.71 (2.75) |  |  |  |
  Day 84 (Week 12) - Negative symptoms: number analyzed (Participants) | 10 | 6 | 31 | 4 | 20 | 21
  Day 84 (Week 12) - Negative symptoms | 18.90 (5.38) | 15.33 (3.08) | 20.5 (5.9) | 22.5 (4.8) | 18.6 (4.4) | 19.4 (4.8)
  Baseline - Positive symptoms: number analyzed (Participants) | 14 | 12 | 37 | 5 | 30 | 32
  Baseline - Positive symptoms | 17.93 (3.99) | 19.75 (3.93) | 18.9 (4.6) | 18.0 (3.7) | 17.6 (4.2) | 17.2 (5.4)
  Day 14 - Positive symptoms: number analyzed (Participants) | 13 | 10 | 36 | 4 | 26 | 30
  Day 14 - Positive symptoms | 18.23 (4.75) | 21.30 (4.35) | 17.8 (3.8) | 18.3 (5.3) | 18.1 (3.9) | 18.0 (5.7)
  Day 28 - Positive symptoms: number analyzed (Participants) | 10 | 9 | 33 | 3 | 26 | 28
  Day 28 - Positive symptoms | 17.60 (4.77) | 19.22 (5.19) | 17.9 (4.3) | 24.3 (6.0) | 18.0 (4.9) | 17.4 (5.9)
  Day 42 - Positive symptoms: number analyzed (Participants) | 11 | 8 | 32 | 4 | 24 | 24
  Day 42 - Positive symptoms | 17.82 (4.31) | 18.75 (4.13) | 18.2 (4.8) | 22.5 (6.0) | 16.0 (4.4) | 16.2 (4.7)
  Day 56 - Positive symptoms: number analyzed (Participants) | 10 | 7 | 33 | 4 | 24 | 23
  Day 56 - Positive symptoms | 17.90 (4.93) | 20.71 (1.50) | 17.7 (5.0) | 20.5 (3.1) | 17.2 (6.1) | 15.8 (4.5)
  Day 70 - Positive symptoms: number analyzed (Participants) | 10 | 7 | 0 | 0 | 0 | 0
  Day 70 - Positive symptoms | 19.20 (2.86) | 19.29 (2.69) |  |  |  |
  Day 84 (Week 12) - Positive symptoms: number analyzed (Participants) | 10 | 6 | 31 | 4 | 20 | 21
  Day 84 (Week 12) - Positive symptoms | 17.70 (5.25) | 19.67 (3.61) | 17.3 (4.5) | 21.5 (2.6) | 16.5 (4.7) | 15.5 (4.3)

8. Secondary Outcome: Brief Negative Symptom Scale (BNSS) Total Scores
Description: The BNSS is a 13-item instrument designed for clinical trials that measures the severity of the negative symptoms of schizophrenia in five domains. There are 13 items organized into 6 subscales (anhedonia, distress, asociality, avolition, blunted affect, and alogia), each rated on a 7-point scale (0-6) where 0 = absent symptoms and 6 = severe symptoms. The total score is calculated by summing the individual items (13) of each subscale and has a range of 0-78.
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part A: Monotherapy (Placebo) | Part A: Monotherapy (150 mg) | Part B: Add-on Therapy (Placebo) | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
Number analyzed (Participants) | 15 | 12 | 37 | 5 | 30 | 32
Units on a scale
  Baseline: number analyzed (Participants) | 14 | 12 | 36 | 5 | 29 | 32
  Baseline | 34.79 (14.98) | 35.17 (13.68) | 36.6 (14.9) | 36.4 (6.7) | 38.1 (13.7) | 38.4 (13.8)
  Day 14: number analyzed (Participants) | 13 | 10 | 36 | 4 | 25 | 30
  Day 14 | 35.08 (12.48) | 32.90 (13.47) | 36.1 (11.4) | 29.3 (11.1) | 34.1 (12.8) | 35.2 (12.8)
  Day 28: number analyzed (Participants) | 10 | 8 | 33 | 3 | 26 | 28
  Day 28 | 29.90 (14.49) | 33.25 (8.94) | 32.6 (12.9) | 32.7 (7.4) | 33.1 (13.4) | 36.5 (10.3)
  Day 42: number analyzed (Participants) | 11 | 8 | 32 | 4 | 24 | 24
  Day 42 | 34.09 (11.95) | 36.38 (14.79) | 35.1 (11.3) | 35.0 (11.8) | 35.5 (12.6) | 32.7 (13.4)
  Day 56: number analyzed (Participants) | 10 | 7 | 31 | 4 | 24 | 23
  Day 56 | 37.40 (18.60) | 34.00 (12.12) | 30.3 (12.1) | 37.5 (16.3) | 30.8 (11.8) | 32.3 (13.6)
  Day 70: number analyzed (Participants) | 10 | 7 | 0 | 0 | 0 | 0
  Day 70 | 33.10 (7.23) | 34.00 (15.15) |  |  |  |
  Day 84 (Week 12): number analyzed (Participants) | 10 | 6 | 31 | 4 | 19 | 21
  Day 84 (Week 12) | 30.40 (12.86) | 28.17 (20.44) | 32.7 (13.4) | 33.3 (10.6) | 29.6 (9.2) | 29.2 (12.4)

9. Secondary Outcome: Defeatist Performance Attitude Scale (DPAS) Scores
Description: The DPAS is a 15-item, patient-rated assessment that evaluates expectations of failures or self-defeating beliefs related to prior failed experiences as well as illness on a 7-point Likert scale (total range = 15-105) ranging from totally agree (1) to totally disagree (7).
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part A: Monotherapy (Placebo) | Part A: Monotherapy (150 mg) | Part B: Add-on Therapy (Placebo) | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
Number analyzed (Participants) | 15 | 12 | 37 | 5 | 30 | 32
Units on a scale
  Baseline | 34.73 (13.92) | 30.25 (12.43) | 40.2 (14.6) | 40.0 (6.4) | 38.2 (15.9) | 35.9 (16.2)
  Day 42: number analyzed (Participants) | 13 | 10 | 32 | 4 | 24 | 26
  Day 42 | 40.54 (16.37) | 27.50 (18.65) | 37.5 (14.2) | 39.3 (9.3) | 38.8 (16.2) | 36.0 (16.2)
  Day 84 (Week 12): number analyzed (Participants) | 10 | 6 | 31 | 4 | 20 | 22
  Day 84 (Week 12) | 38.80 (13.42) | 16.00 (4.98) | 36.0 (15.2) | 54.3 (16.4) | 39.0 (19.9) | 32.2 (13.6)

10. Secondary Outcome: Number of Participants With Suicidal Ideation or Behavior, and Self-injurious Behavior Without Suicidal Intent on the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a suicide risk assessment tool used to help identify the risk of suicide.
Time Frame: Baseline through Day 84
Population: The safety population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Number of participants
Arm/Group | Part A: Monotherapy (Placebo) | Part A: Monotherapy (150 mg) | Part B: Add-on Therapy (Placebo) | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
Number analyzed (Participants) | 15 | 12 | 37 | 5 | 30 | 32
Number of participants
  Suicidal ideation or behavior | 0 | 0 | 1 | 0 | 2 | 1
  Self-injurious behavior without suicidal intent | 1 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Extrapyramidal Symptom Rating Scale, Abbreviated (ESRS-A)
Description: The ESRS-A is used to evaluate the presence and severity of extrapyramidal symptoms. Items are rated on a scale of 0 (no symptoms) to 5 (extreme symptoms).
Time Frame: Baseline through Day 84
Population: The safety population included all randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part A: Monotherapy (Placebo) | Part A: Monotherapy (150 mg) | Part B: Add-on Therapy (Placebo) | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
Number analyzed (Participants) | 15 | 12 | 37 | 5 | 30 | 32
Units on a scale
  Akathisia Baseline: number analyzed (Participants) | 15 | 12 | 37 | 4 | 30 | 32
  Akathisia Baseline | 0.07 (0.26) | 0.08 (0.29) | 0.27 (0.87) | 0.00 (0.00) | 0.27 (0.83) | 0.38 (0.98)
  Akathisia Day 84: number analyzed (Participants) | 10 | 6 | 31 | 3 | 20 | 21
  Akathisia Day 84 | 0.00 (0.00) | 0.00 (0.00) | 0.29 (0.94) | 0.00 (0.00) | 0.10 (0.45) | 0.10 (0.44)
  Dyskinesia Baseline: number analyzed (Participants) | 15 | 12 | 37 | 4 | 30 | 32
  Dyskinesia Baseline | 0.00 (0.00) | 0.33 (0.89) | 0.46 (1.95) | 0.75 (0.96) | 0.17 (0.38) | 0.63 (1.68)
  Dyskinesia Day 84: number analyzed (Participants) | 10 | 6 | 31 | 3 | 20 | 21
  Dyskinesia Day 84 | 0.10 (0.32) | 0.00 (0.00) | 0.16 (0.90) | 0.00 (0.00) | 0.15 (0.49) | 0.29 (0.72)
  Dystonia Baseline | 0.07 (0.26) | 0.00 (0.00) | 0.24 (0.86) | 0.00 (0.00) | 0.03 (0.18) | 0.16 (0.51)
  Dystonia Day 84: number analyzed (Participants) | 10 | 6 | 31 | 3 | 20 | 21
  Dystonia Day 84 | 0.00 (0.00) | 0.00 (0.00) | 0.26 (1.03) | 0.00 (0.00) | 0.05 (0.22) | 0.00 (0.00)
  Parkinsonism Baseline | 0.13 (0.52) | 0.42 (1.00) | 1.03 (2.36) | 2.20 (1.92) | 2.00 (3.24) | 2.22 (4.15)
  Parkinsonism Day 84: number analyzed (Participants) | 10 | 6 | 31 | 3 | 20 | 21
  Parkinsonism Day 84 | 0.20 (0.63) | 0.33 (0.82) | 1.03 (2.87) | 0.33 (0.58) | 1.15 (2.68) | 1.00 (2.30)

12. Secondary Outcome: Maximum Serum Concentration (Cmax) of RO6889450
Time Frame: Day 42
Population: The pharmacokinetic population consisted of all participants who received at least one dose of study drug and who had data from at least one post-dose sample. It was pre-specified to not summarize and report Part A PK data, which was used only for model building.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
Number analyzed (Participants) | 4 | 27 | 28
ng/mL | 157 (58.7) | 794 (40.3) | 1550 (43.9)

13. Secondary Outcome: Area Under the Curve at Steady State (AUCss) of RO6889450
Time Frame: Day 42
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
Number analyzed (Participants) | 4 | 27 | 28
h*ng/mL | 2980 (54.8) | 15100 (43.8) | 28600 (48.4)

ADVERSE EVENTS:
Time Frame: Up to Day 84 (Week 12)
Arm/Group | Part A: Monotherapy (Placebo) | Part A: Monotherapy (150 mg) | Part B: Add-on Therapy (Placebo) | Part B: Add-on Therapy (45 mg) | Part B: Add-on Therapy (150 mg) | Part B: Add-on Therapy (300 mg)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/12 | 1/37 | 0/5 | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/12 | 1/37 | 0/5 | 2/30 | 0/32
Other Adverse Events (participants affected / at risk) | 7/15 | 4/12 | 9/37 | 2/5 | 8/30 | 4/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Monotherapy (Placebo) (N=15) | Part A: Monotherapy (150 mg) (N=12) | Part B: Add-on Therapy (Placebo) (N=37) | Part B: Add-on Therapy (45 mg) (N=5) | Part B: Add-on Therapy (150 mg) (N=30) | Part B: Add-on Therapy (300 mg) (N=32)
Accidental death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Monotherapy (Placebo) (N=15) | Part A: Monotherapy (150 mg) (N=12) | Part B: Add-on Therapy (Placebo) (N=37) | Part B: Add-on Therapy (45 mg) (N=5) | Part B: Add-on Therapy (150 mg) (N=30) | Part B: Add-on Therapy (300 mg) (N=32)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT03669640/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT03669640/SAP_001.pdf